CLINICAL TRIAL: NCT02709915
Title: Effect of Meal Frequency and Timing on Glycemic Control, Daily Insulin Dose Requirements and Clock Gene Expression in Uncontrolled Type 2 Diabetic Patients
Brief Title: Effect of Meal Frequency and Timing on Insulin Dose and Clock Gene in Type 2 Diabetic Patients
Acronym: Bdiet-6Mdiet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Daniela Jakubowicz, Professor, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0233-15-WOMC
Record Dates: First submitted 2016-03-07; First posted 2016-03-16 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breakfast Diet (Bdiet) (Experimental): The Bdiet will consist in 3 meals with distribution of calories: breakfast 50%, lunch 33% and dinner 17%.
  Interventions: Other: Breakfast Diet (Bdiet); Other: 6Meal Diet (6Mdiet
- 6 small meals diet (6Mdiet) (Active Comparator): The 6Mdiet will consist on 6 meals (breakfast, lunch and dinner and 3 snacks) with distribution of calories: breakfast 15%, lunch 25%, dinner 30% and 10% each of the three snacks.
  Interventions: Other: Breakfast Diet (Bdiet); Other: 6Meal Diet (6Mdiet

INTERVENTIONS:
Other: Breakfast Diet (Bdiet) — The Breakfast Ddiet consist of high-energy breakfast, medium-sized lunch and reduced in energy dinner, with distribution of calories: breakfast 50%, lunch 33% and dinner 17%. In this diet, the investigators will evaluate at baseline and at the end of 12 weeks of diet intervention, the diet efficacy on reducing HbA1c, the total daily insulin dose requirements (TDID), the efficacy on reducing body weight, fasting plasma glucose (FPG) and overall glycemic excursion assessed with continuous monitoring system. The investigators will assess also the Clock Genes mRNA expression in white blood cells. at baseline and after 12 weeks of diet intervention
  Other Names: Bdiet
Other: 6Meal Diet (6Mdiet — The 6meal diet (6Mdiet) will consist in the traditional antidiabetic diet, consuming 6 small meals: breakfast, lunch and dinner and 3 snacks, with caloric distribution: breakfast 20%, lunch 25%, dinner 25% and 10% each of the 3 snacks. In this diet, the investigators will evaluate at the beginning and at the end of the study (12 weeks), the diet effects on reducing HbA1c, total daily insulin dose requirements (TDID), and the diet efficacy on reducing body weight, fasting plasma glucose (FPG) and overall glycemic excursion, using continuous monitoring system, The investigators will assess also at baseline and at the end of the diet intervention the Clock Genes mRNA expression in white blood cells.
  Other Names: 6Mdiet

SUMMARY:
This study is undertaken to explore in patients with uncontrolled T2D treated with insulin, whether a diet with large breakfast and lunch with small dinner (Bdiet) will enhance CG expression and will be more effective for weight loss and for achieving glycemic control and reduction of total daily insulin dose (first end point), compared to an isocaloric diet with 6 small meals distributed evenly along the day

DETAILED DESCRIPTION:
Obese patients with type 2 diabetes (T2D) and insulin resistance (IR), often require sequential increments of total daily insulin dose (TDID). This causes weight gain, worsens IR, leading to further increase of TDID and persistent hyperglycemia. In these patients, weight loss (WL) and reduction of IR are mandatory in order to achieve glucose control with less TDID. Impaired clock gene (CG) expression is linked to obesity and IR in T2D and it was shown in animals and T2D patients treated with oral anti-hyperglycemic drugs, that WL diet with restricted meal timing to specific hours, restored CG expression and was more effective for WL and for reduction of hyperglycemia compared to isocaloric WL diet, (commonly recommended for T2D), consisting of small meals randomly distributed along the day.

The investigators hypothesized that in patients with uncontrolled T2D treated with insulin, a diet with large breakfast and lunch with small dinner (Bdiet) will enhance CG expression and will be more effective for WL and for achieving glycemic control and reduction of TDID, compared to an isocaloric diet with 6 small meals distributed evenly along the day (6Mdiet).

This will be a randomized parallel, open label clinical study. Thirty overweight and obese insulin-treated T2D patients with HbA1c>7.5% will be assigned to 12 weeks of 2 isocaloric diets: either Bdiet or 6Mdiet. HbA1c and CG mRNA expression in white blood cells and overall daily glycemia measured during 14 days, will be assessed before diet, after 14 days and at the end of the diet intervention. The TDID (first end point ) will be adjusted by physician, according to the results of self-monitoring of blood glucose on 3 consecutive days at baseline and before each of the visits.

ELIGIBILITY:
Inclusion Criteria:

* T2D patients with stable insulin treatment for at least 3 month preceding the study.
* HgA1c >7.5 %.
* Age > 30 years.
* BMI: 27-34 kg/m2.
* Treatment with antidiabetic drugs (i.e. metformin, DPP4 inhibitors, glinides) and GLP-1 analogs.
* Anti-hypertensive treatment will be allowed.
* Lipid-lowering medication.

Exclusion Criteria

* Type 1 diabetes.
* Major illnesses (liver, heart, kidney, infectious, neurological, psychiatric, immunological, active malignancy).
* Presently dieting.
* Change in weight of > 4.5 kg within 3 month prior to study onset.
* Night or rotating shift workers.
* Those who crossed more than 2 time zones during 2-week period prior to study onset.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Insulin Dose | Baseline, 2 week and at 12 weeks
  The effects of two diets (Bdiet and 6Mdiet) will be compared on their efficacy on total insulin dose reduction measured at baseline, after 2 weeks and at the end (12 weeks) of both diet interventions

SECONDARY OUTCOMES:
HbA1c | Baseline, 2 weeks and at 12 weeks
  The effect of the two diets (Bdiet and 6Mdiet) will be compared on the efficacy on the reduction of HbA1c measured at baseline, after 2 weeks and at the end (12 weeks) of both diet interventions
Overall Glycemia | Baseline, 2 week and at 12 weeks
  The effect of the two diets on all-day glycemia will be assessed with continuous blood monitoring system at baseline, after 2 weeks and after 12 weeks of the two diet intervention
Clock Gene mRNA expression | Baseline, 2 week and at 12 weeks
  The measurement of mRNA expression of clock gene in circulating white blood cells will be assessed at baseline, after 2 weeks and after 12 weeks of the two diet intervention

OTHER OUTCOMES:
Body Weight | Baseline, 2 week and at 12 weeks
  The measurement of body weight assessed at baseline, after 2 weeks and after 12 weeks of the two diet intervention

CONTACTS AND LOCATIONS:
Overall Officials: Julio Wainstein, MD, Principal Investigator — Wolfson Medical Center
Locations (1):
- Daniela Jakubowicz, Holon, Wolfson Medical Center, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jakubowicz D, Landau Z, Tsameret S, Wainstein J, Raz I, Ahren B, Chapnik N, Barnea M, Ganz T, Menaged M, Mor N, Bar-Dayan Y, Froy O. Reduction in Glycated Hemoglobin and Daily Insulin Dose Alongside Circadian Clock Upregulation in Patients With Type 2 Diabetes Consuming a Three-Meal Diet: A Randomized Clinical Trial. Diabetes Care. 2019 Dec;42(12):2171-2180. doi: 10.2337/dc19-1142. Epub 2019 Sep 23. PMID 31548244